CLINICAL TRIAL: NCT00853866
Title: Entwicklung Neuronaler Repräsentationen Nach Schlaganfall: Verbesserung Motorischer Leistungen Durch Transkranielle Gleichstromstimulation Und Noradrenerge Co-Stimulation
Brief Title: Enhancement of Motor Function with Reboxetine and Transcranial Direct Current Stimulation
Acronym: STIMBOX
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: German Research Foundation (Other); University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2005-00160436-36; 28/2005AMG1 (Other: AMG); SFB550 TPC5 (Other: Deutsche Forschungsgemeinschaft (DFG))
Record Dates: First submitted 2009-02-27; First posted 2009-03-02 (Estimated); Last update posted 2024-12-10 (Actual); Status verified 2017-08

CONDITIONS: Cerebral Stroke
Keywords: stroke; reboxetine; noradrenaline; motor cortex; transcranial direct current stimulation; motor function; rehabilitation; Jebsen Taylor test
MeSH Terms: conditions — Stroke | interventions — Reboxetine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- RBX + tDCS (Experimental): reboxetine + tDCS verum
  Interventions: Drug: reboxetine; Device: tDCS verum
- RBX + sham stimulation (Active Comparator): reboxetine + sham tDCS
  Interventions: Drug: reboxetine; Device: tDCS sham
- PLC + tDCS (Active Comparator): placebo drug + verum tDCS
  Interventions: Drug: Placebo; Device: tDCS verum
- PLC + sham stimulation (Sham Comparator): placebo drug + sham tDCS
  Interventions: Drug: Placebo; Device: tDCS sham

INTERVENTIONS:
Drug: reboxetine — single dose of 4mg reboxetine 80 minutes before assessment of Jebsen Taylor test
  Other Names: brand name: Edronax, serial number: KPR 08092410/11
  Arms: RBX + sham stimulation; RBX + tDCS
Drug: Placebo — placebo, 80 min before assessment of Jebsen Taylor test
  Other Names: placebo drug resembling Edronax
  Arms: PLC + sham stimulation; PLC + tDCS
Device: tDCS verum — 20 minutes of 1 mV transcranial direct current stimulation with 5x5 cm electrodes with active electrode over the primary motor representation of the stroke hemisphere and reference electrode over the contralateral supraorbital area Application during assessment of Jebsen Taylor test
  Other Names: Hersteller:; DC Stimulator; Manufacturer:; eldith -Electro-Diagnostic & Therapeutic Systems GmbH; Gustav-Kirchhoff-Straße 5; D-98693 Ilmenau; Serialnumber: 0006
  Arms: PLC + tDCS; RBX + tDCS
Device: tDCS sham — 30 seconds of 1 mV transcranial direct current stimulation with 5x5 cm electrodes with active electrode over the primary motor representation of the stroke hemisphere and reference electrode over the contralateral supraorbital area Application during assessment of Jebsen Taylor test
  Other Names: Hersteller:; DC Stimulator; Manufacturer:; eldith -Electro-Diagnostic & Therapeutic Systems GmbH; Gustav-Kirchhoff-Straße 5; D-98693 Ilmenau; Serialnumber: 0006
  Arms: PLC + sham stimulation; RBX + sham stimulation

SUMMARY:
The hypothesis of the study is that combination of reboxetine/tDCS is more effective in enhancing motor functions of daily life (assessed by the Jebsen Taylor test) as compared to reboxetine and tDCS alone. The protocol is designed as a within-subject, block randomized placebo-controlled double-blind crossover study.

DETAILED DESCRIPTION:
One important feature of the human brain is the ability to undergo plastic changes and reorganization after learning and lesions of the nervous system. This ability is of major importance for the treatment of functional deficits after stroke. Stroke is the major disease leading to persistent functional disabilities in Germany. However, the success rate of therapeutic interventions, especially in chronic stroke patients, is still unsatisfactory. Thus, basic science is essential to discover new therapeutic options that bear the potential for translation into clinical practice. Recent evidence is pointing to modulating the motor cortical excitability in order to enhance motor function in stroke patients. For this purpose, reboxetine as a selective reuptake inhibitor of noradrenaline and transcranial direct current stimulation have proven effective in enhancing motor functions needed for daily life activities by 10-12%. These improvements were significant compared to placebo, but still clinically unsatisfactory. Thus, this protocol aims at enhancing the excitability modulatory effect of each single intervention through the combination of reboxetine and tDCS. The hypothesis of the study is that combination of reboxetine/tDCS is more effective in enhancing motor functions of daily life (assessed by the Jebsen Taylor test) as compared to reboxetine and tDCS alone.

The protocol is designed as a within-subject, block randomized placebo-controlled double-blind crossover study. 12 chronic stroke patients with persistent functional deficits of the arm and/or hand will be included. The primary outcome measure is the time needed to fulfill all subtests of the Jebsen Taylor test. All patients undergo four different conditions in four different sessions: 1) reboxetine + verum tDCS; 2) reboxetine + sham tDCS 3) placebo drug + verum tDCS 4) placebo drug + sham tDCS.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 86
* patient is contractually capable
* first-ever, ischemic stroke
* minimum time since stroke 9 months
* a paresis of the arm/hand muscles above 3 on the MRC scale

Exclusion Criteria:

* multiple cerebral lesions and associated residual deficits
* severe head trauma in the past
* seizures
* ferromagnetic implants in the head/neck region
* pacemaker
* a psychiatric disorder or neurological disease besides stroke
* intake of illegal drugs
* severe aphasia or cognitive deficits that impede contractual capability
* contraindications for reboxetine (seizures, glaucoma, prostate hyperplasia with urinary retention, cardiac arrhythmias, potential interactions with co-medication)
* pregnancy
* breast-feeding patients

Ages: 18 Years to 86 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-01; Primary Completion 2009-11 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
JTT | crossover design, four different sessions with four different interventions
  Jebsen Taylor test

SECONDARY OUTCOMES:
Force | crossover design, four different sessions with four different interventions
  maximum grip force
NHPT | crossover design, four different sessions with four different interventions
  nine hole peg test

CONTACTS AND LOCATIONS:
Overall Officials: Christian Gerloff, MD, Principal Investigator — Department of Neurology, University Hospital Hamburg-Eppendorf
Locations (1):
- University Hospital Hamburg-Eppendorf, Department of Neurology, Hamburg, Hamburg, Germany

REFERENCES:
- [Background] Hummel F, Celnik P, Giraux P, Floel A, Wu WH, Gerloff C, Cohen LG. Effects of non-invasive cortical stimulation on skilled motor function in chronic stroke. Brain. 2005 Mar;128(Pt 3):490-9. doi: 10.1093/brain/awh369. Epub 2005 Jan 5. PMID 15634731
- [Background] Hummel F, Cohen LG. Improvement of motor function with noninvasive cortical stimulation in a patient with chronic stroke. Neurorehabil Neural Repair. 2005 Mar;19(1):14-9. doi: 10.1177/1545968304272698. PMID 15673839
- [Background] Hummel FC, Voller B, Celnik P, Floel A, Giraux P, Gerloff C, Cohen LG. Effects of brain polarization on reaction times and pinch force in chronic stroke. BMC Neurosci. 2006 Nov 3;7:73. doi: 10.1186/1471-2202-7-73. PMID 17083730
- [Background] Plewnia C, Hoppe J, Gerloff C. No effects of enhanced central norepinephrine on finger-sequence learning and attention. Psychopharmacology (Berl). 2006 Aug;187(2):260-5. doi: 10.1007/s00213-006-0420-5. Epub 2006 Jun 10. PMID 16767410
- [Background] Plewnia C, Hoppe J, Cohen LG, Gerloff C. Improved motor skill acquisition after selective stimulation of central norepinephrine. Neurology. 2004 Jun 8;62(11):2124-6. doi: 10.1212/01.wnl.0000128041.92710.17. PMID 15184632
- [Background] Plewnia C, Hoppe J, Hiemke C, Bartels M, Cohen LG, Gerloff C. Enhancement of human cortico-motoneuronal excitability by the selective norepinephrine reuptake inhibitor reboxetine. Neurosci Lett. 2002 Sep 27;330(3):231-4. doi: 10.1016/s0304-3940(02)00803-0. PMID 12270635
- [Derived] Elsner B, Kugler J, Pohl M, Mehrholz J. Transcranial direct current stimulation (tDCS) for improving activities of daily living, and physical and cognitive functioning, in people after stroke. Cochrane Database Syst Rev. 2020 Nov 11;11(11):CD009645. doi: 10.1002/14651858.CD009645.pub4. PMID 33175411
- See also: Homepage Brain Imaging and Neurostimulation Lab, Department of Neurology, University Hospital Hamburg-Eppendorf — https://www.uke.de/english/departments-institutes/departments/neurology/research/index.html